CLINICAL TRIAL: NCT04070378
Title: An Open-Label, Pilot Study of Daratumumab SC in Patients With Mild to Moderate Alzheimer's Disease
Brief Title: Study of Daratumumab in Patients With Mild to Moderate Alzheimer's Disease
Acronym: DARZAD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Marc L Gordon, MD (Other)
Collaborators: Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Sponsor-Investigator, Marc L Gordon, MD, Professor of Neurology and Psychiatry, Northwell Health
Organization: Northwell Health (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-0619
Record Dates: First submitted 2019-08-22; First posted 2019-08-28 (Actual); Results first posted 2023-11-29 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2023-11

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — daratumumab

STUDY DESIGN:
Intervention Model Description: Open-label treatment group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open-label Treatment (Experimental): This is an open-label pilot study designed to explore whether daratumumab may have a clinically meaningful effect in patients with mild to moderate Alzheimer's disease. During the treatment phase, eligible subjects will receive daratumumab SC 1800 mg (daratumumab 1800 mg with rHuPH20 30,000 units) subcutaneous infusion over 3-5 minutes (15 mL) once weekly for 8 weeks followed by daratumumab SC 1800 mg every 2 weeks for 16 weeks.
  Interventions: Drug: Daratumumab Injection

INTERVENTIONS:
Drug: Daratumumab Injection — Daratumumab SC 1800 mg (daratumumab 1800 mg with rHuPH20 30,000 units) subcutaneous infusion

SUMMARY:
This is an open-label, pilot study designed to explore whether daratumumab may have a clinically meaningful effect in patients with mild to moderate Alzheimer's disease.

DETAILED DESCRIPTION:
Daratumumab is a human antibody that targets CD38. It is FDA-approved for the treatment of multiple myeloma, has broad-ranging immunomodulatory effects on nonplasma cells that express CD38, and is able to cross the blood-brain barrier. CD38 expression on CD8+ T-cells is significantly increased in the blood of early AD patients as compared with age-matched controls, and activated T-cells are capable of trafficking into the central nervous system and exerting toxic effects. This study is designed to explore whether treatment with Daratumumab may have a clinically meaningful effect on patients with mild to moderate Alzheimer's disease.

ELIGIBILITY:
Inclusion Criteria:

1. Each subject must be ≥ 55 to ≤ 85 years of age at the screening visit.
2. Each subject must have a diagnosis of probable AD dementia according to National Institute on Aging-Alzheimer's Association (NIA-AA) criteria.
3. Each subject must have a Mini-Mental State Examination (MMSE) score ≥ 15 and ≤ 26 at the screening visit.
4. Each subject must have a Magnetic Resonance Imaging (MRI) scan performed during the screening period that is consistent with a diagnosis of AD.
5. Each subject must have a positive amyloid Positron Emission Tomography (PET) scan, either performed during the screening period, or previously performed provided that the scan and result are considered acceptable by the investigator.
6. If the subject is receiving a cholinesterase inhibitor (donepezil, rivastigmine, or galantamine) and/or memantine, the dose must have been stable for at least 12 weeks before the screening visit, and the subject must be willing to remain on the same dose for the duration of the trial.
7. Each subject must have a study partner who is reliable and competent. The study partner must have a close relationship with the subject, have face to face contact at least 3 days/week for a minimum of 6 waking hours/week, and be willing to accompany the subject to all required study visits.
8. Each subject must have no clinically significant abnormal laboratory test results [complete blood count (CBC), prothrombin time (PT)/international normalized ratio (INR), activated partial thromboplastin time (APTT), comprehensive metabolic panel (CMP), thyroid stimulating hormone (TSH), and vitamin B12 level] at the screening visit.
9. Each subject must have results of a physical and neurological examination and vital signs within normal limits or clinically acceptable to the investigator at the screening visit.
10. If female, the subject must be postmenopausal defined as: No menses for 12 or more months without an alternative medical cause OR permanently surgically sterile (bilateral oophorectomy, bilateral salpingectomy, or hysterectomy).

Exclusion Criteria:

1. The subject has a Rosen-modified Hachinski Ischemia Score > 4 at the screening visit.
2. The subject has a known history of stroke or evidence from screening MRI that is clinically significant in the investigator's opinion.
3. The subject has evidence of a clinically relevant neurological disorder other than probable AD at the screening visit, including: vascular dementia, Parkinson's disease, dementia with Lewy bodies, frontotemporal dementia, progressive supranuclear palsy, corticobasal degeneration, amyotrophic lateral sclerosis, Huntington's disease, multiple sclerosis, mental retardation, hypoxic cerebral damage, or head trauma with loss of consciousness that led to persistent cognitive deficits.
4. The subject has evidence of a clinically relevant or unstable psychiatric disorder, based on DSM-5 criteria, including schizophrenia or other psychotic disorder, bipolar disorder, delirium, or major depression. (Major depression in remission is not exclusionary.) A score on the 15-item Geriatric Depression Scale (GDS) of 5 or more requires an assessment by an appropriate health care professional to evaluate for the presence of major depression. Subjects with a score of 5 or more who are not diagnosed with major depression following such an assessment may be included in the trial.
5. The subject has a history of alcoholism or drug dependency/abuse within the last 5 years before screening.
6. The subject has been treated with any investigational product within 60 days or 5 half-lives (whichever is longer) prior to the screening visit.
7. The subject has been treated with anti-amyloid-beta or anti-tau protein monoclonal antibodies within one year prior to the screening visit.
8. The subject has been treated with an active vaccine targeting amyloid-beta or tau protein.
9. The subject has received a live/live-attenuated bacterial or viral vaccine within 3 months prior to the screening visit.
10. The subject has been treated with immunosuppressive medications, such as azathioprine, cyclosporine, methotrexate, tacrolimus, or mycophenylate, within 2 months prior to the screening visit.
11. The subject has been treated with a course of corticosteroids longer than 5 days within 2 months prior to the screening visit.
12. The subject is taking or is anticipated to require treatment with estrogens.
13. The subject is taking or is anticipated to require treatment with an anticoagulant medication, including warfarin, dabigatran, rivaroxaban, apixaban, edoxaban, heparin, or enoxaparin.
14. The subject is taking or is anticipated to require treatment with aspirin at a dose higher than 325 mg daily.
15. The subject has a history of asthma or chronic obstructive pulmonary disease.
16. The subject has had a myocardial infarction, unstable angina, stroke, transient ischemic attack or required intervention for any of these conditions (e.g., coronary artery bypass graft, percutaneous coronary intervention via cardiac catheterization, thrombolytic therapy) within 6 months prior to the screening visit.
17. The subject has had an infection requiring medical intervention within 30 days prior to the screening visit.
18. The subject has serologic evidence of current or prior hepatitis B virus (HBV) infection based on hepatitis B surface antigen or hepatitis core antibody blood tests at the screening visit.
19. The subject has serologic evidence of hepatitis C virus (HCV) infection based on hepatitis C antibody blood test at the screening visit.
20. The subject has serologic evidence of human immunodeficiency virus (HIV) infection based on HIV antigen/antibody test at the screening visit.
21. The subject has a platelet count less than 50,000 per microliter (mL) at the screening visit.
22. The subject has a creatinine clearance less than 30 mL/minute at the screening visit.
23. The subject has a history or evidence of a malignancy (except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or localized prostate carcinoma) within the 2 years prior to the screening visit.
24. The subject has had any other unstable/uncontrolled medical illness within 12 weeks prior to the screening visit such that, in the judgment of the investigator, participation in the trial would pose a significant medical risk to the subject.
25. The subject has significant visual or auditory impairment, or limited English proficiency, that in the investigator's opinion would preclude collection of outcome measures.
26. The subject has any contraindication to or inability to tolerate brain MRIs (e.g., a pacemaker or any other implanted device or condition that would preclude proximity to a strong magnetic field).
27. The subject has any contraindication to or inability to tolerate a PET scan (includes current or recent participation in any procedures involving radioactive agents such that the total radiation dose exposure to the subject in any given year would exceed acceptable limits of annual and total dose).
28. The subject has a history of allergy to dexamethasone, diphenhydramine, acetaminophen, montelukast, or acyclovir.

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2019-11-06 (Actual); Primary Completion 2023-06-08 (Actual); Study Completion 2023-08-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The Litwin-Zucker Research Center, Manhasset, New York, United States

IPD SHARING:
Plan to Share IPD: No
This study will comply with the Clinical Trials Registration and Results Information Submission rule. Result information from this trial will be submitted to ClinicalTrials.gov.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Open-label Treatment
Started | 16
Subjects who received at least one dose of study drug. | 9
Completed | 6
Not Completed | 10
Not completed — Withdrawal by Subject | 2
Not completed — Screen Failure | 6
Not completed — Physician Decision | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Open-label Treatment
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 10
Age, Continuous [Mean (Full Range); unit: years] | 67.46 [55.75 to 80.38]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 13
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With an Improvement of ≥ 4 Points on the ADAS-cog/11
Description: The standard 11-item version of the Alzheimer's Disease Assessment Scale, cognitive subscale score (ADAS-cog/11) includes both subject-completed tests and observer-based assessments. Specific tasks include Word Recall, Naming Objects and Fingers, Commands, Constructional Praxis, Ideational Praxis, Orientation, Word Recognition, and Language. The score ranges from 0 to 70 with each point representing a performance error and higher scores reflecting worse performance. An improvement (decrease) of ≥ 4 points in ADAS-cog/11 score has been deemed to be clinically meaningful.
Time Frame: 25 weeks
Population: A total of 16 subjects were screened, with 6 screen failures, 1 subject who withdrew consent prior to treatment, 1 subject who withdrew consent after 3 treatment visits, 1 subject withdrawn by the investigator after having missed 7 consecutive visits due to the COVID pandemic, and 1 subject withdrawn due to a possibly related adverse event, leaving 6 evaluable subjects who completed treatment.
Measure: Number; unit: responders
Arm/Group | Open-label Treatment
Number analyzed (Participants) | 6
responders | 0

2. Secondary Outcome: The Number of Subjects Who Are Unchanged or Improved From Baseline on ADAS-cog/12 Score
Description: The 12-item version of the Alzheimer's Disease Assessment Scale, cognitive subscale (ADAS-Cog/12) adds a delayed word recall task, scored from 0 to 10. The ADAS-Cog/12 score is the total of the ADAS-Cog/11 plus the delayed recall score, and therefore has a range of 0 to 80. Higher scores reflect worse performance.
Time Frame: 25 weeks
Population: as for outcome 1
Measure: Number; unit: responders
Arm/Group | Open-label Treatment
Number analyzed (Participants) | 6
responders | 0

3. Secondary Outcome: The Number of Subjects Who Are Unchanged or Improved From Baseline on the MMSE
Description: The Mini-Mental State Examination (MMSE) is a 30-point scale that measures orientation to time and place, registration, immediate and delayed recall, attention, language, and drawing. Scores range from 0 (most impaired) to 30 (no impairment).
Time Frame: 25 weeks
Population: as for outcome 1
Measure: Number; unit: responders
Arm/Group | Open-label Treatment
Number analyzed (Participants) | 6
responders | 0

4. Secondary Outcome: The Number of Subjects Who Are Unchanged or Improved From Baseline on the CDR-SB
Description: The Clinical Dementia Rating Scale Sum of Boxes (CDR-SB) is a clinical global rating scale requiring the interviewing of both the subject and a study partner who knows and has contact with the subject. The CDR-SB is a clinician-directed assessment of both cognition and function, and is intended to capture the state and therefore the disease stage of the individual. The range of scores is from 0-18, with higher scores being worse.
Time Frame: 25 weeks
Population: as for outcome 1
Measure: Number; unit: responders
Arm/Group | Open-label Treatment
Number analyzed (Participants) | 6
responders | 0

5. Secondary Outcome: The Number of Subjects Who Are Unchanged or Improved From Baseline on the ADCOMS
Description: The AD Composite Score (ADCOMS) is derived from a weighted combination of selected items from the ADAS-cog/12, MMSE, and CDR-SB. The range of the ADCOMS is between 0 and 1.97. A higher score is indicative of greater impairment.
Time Frame: 25 weeks
Population: as for outcome 1
Measure: Number; unit: responders
Arm/Group | Open-label Treatment
Number analyzed (Participants) | 6
responders | 0

6. Secondary Outcome: Treatment Emergent Adverse Effects
Description: The proportion of subjects with treatment-emergent adverse effects from initial treatment through final follow-up study visit.
Time Frame: 35 weeks
Population: Nine participants were treated with study medication. Four subjects experienced adverse events that were either definitely or possibly attributed to the medication by the investigator.
Measure: Count of Participants; unit: Participants
Arm/Group | Open-label Treatment
Number analyzed (Participants) | 9
Participants | 4

7. Secondary Outcome: Treatment Emergent Serious Adverse Effects
Description: The proportion of subjects with treatment-emergent serious adverse effects from initial treatment through final follow-up study visit.
Time Frame: 35 weeks
Population: Nine subjects received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Open-label Treatment
Number analyzed (Participants) | 9
Participants | 1

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from the time of consent through completion of the final study follow-up visit (approximately 10 months).
Arm/Group | Open-label Treatment
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 1/9
Other Adverse Events (participants affected / at risk) | 7/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open-label Treatment (N=9)
COVID-19 pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open-label Treatment (N=9)
Infusion reaction; urticarial rash (Skin and subcutaneous tissue disorders) | 4 (4)
cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bilateral cheek, ear, chin erythematous hives with mild swelling and itching (Skin and subcutaneous tissue disorders) | 1 (1)
Brief transient unresponsiveness (Nervous system disorders) | 1 (2)
Burn on lower back (Skin and subcutaneous tissue disorders) | 1 (1) — Related to use of heating pad for back pain.
Vaccine reaction (Immune system disorders) | 1 (1)
diarrhea (Gastrointestinal disorders) | 2 (2)
Difficulty breathing (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dog bite (Skin and subcutaneous tissue disorders) | 1 (1)
Elevated Liver Transaminases (Hepatobiliary disorders) | 1 (1)
Increased agitation (Psychiatric disorders) | 1 (1)
Fall (General disorders) | 1 (1)
fever (Infections and infestations) | 1 (1)
Floaters (Eye disorders) | 1 (1)
Headache (General disorders) | 4 (12)
Increased sleepiness (General disorders) | 1 (1)
Insomnia (General disorders) | 1 (1)
Intermittent palpitations (Cardiac disorders) | 1 (1)
Intermittent nausea/upset stomach (Gastrointestinal disorders) | 1 (2)
Overactive bladder (Renal and urinary disorders) | 1 (1)
Lower back pain/pull (Musculoskeletal and connective tissue disorders) | 1 (1)
Repetitive sneezing (General disorders) | 1 (1)
Runny nose/itchy eyes (General disorders) | 1 (1) — Allergic response
Scratchy throat (General disorders) | 1 (1) — Allergic response
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
UTI (Renal and urinary disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 7 (10)
Weight loss (General disorders) | 1 (1) — >10% of baseline body weight

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-25): https://cdn.clinicaltrials.gov/large-docs/78/NCT04070378/Prot_SAP_000.pdf